CLINICAL TRIAL: NCT06123130
Title: Clinical Validation of the AIMIGo 12 Lead ECG Synthesis Software for Arrhythmia Detection: A Prospective Multicenter Pivotal Study
Brief Title: AIMIGo 12L ECG Synthesis Software Pivotal Study for Arrythmia Detection
Acronym: VALID-ECG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HeartBeam, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HB-VECG-001
Record Dates: First submitted 2023-11-05; First posted 2023-11-08 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Arrhythmias, Cardiac; Atrial Fibrillation; Atrial Flutter; Bradycardia; Tachycardia
Keywords: Telemedicine; Cardiac Arrhythmia; ECG; Synthesis Software; Diagnostic; Vectorcardiography; Remote Monitoring
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation; Atrial Flutter; Bradycardia; Tachycardia; Disease | interventions — Vectorcardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single Arm (Experimental): The study is a prospective single-arm multicenter clinical trial. Adult patients will be consented and enrolled in an outpatient cardiology office or Arrhythmia Clinic.
  Interventions: Device: Vectorcardiography (VECG)

INTERVENTIONS:
Device: Vectorcardiography (VECG) — Patients enrolled will undergo diagnostic ECG recording: three sets of simultaneous 30s recordings with the investigational device AIMIGo and a standard 12L ECG.
  Other Names: HeartBeam AIMIGo VECG System

SUMMARY:
The study is a prospective single-arm multicenter clinical trial. Adult patients will be consented and enrolled in an outpatient cardiology office or Arrhythmia Clinics.

DETAILED DESCRIPTION:
The purpose of this study is to conduct clinical validation of the AIMIGo 12-lead Synthesis Software against a standard FDA-cleared 12-lead ECG system, based on quantitative and qualitative assessment of paired recordings from the same patient, in sinus rhythm or during episodes of symptomatic non-life-threatening arrhythmia. The study will provide the necessary data for an FDA 510(k) regulatory submission and develop experience for market access and integration into clinical workflows.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects over 18 years of age.
2. Referred to outpatient arrhythmia clinic with a history of one or more of the following conditions:

   1. Previous diagnosis of arrhythmia presenting to the clinic for routine follow-up evaluation.
   2. Patients with symptoms indicative of cardiac arrhythmias.
3. Able and willing to sign informed consent.

Exclusion Criteria:

1. Open chest wounds or recent (<30 days) surgery to the chest or abdomen.
2. Clinical conditions that in the opinion of the Investigator would compromise the safety of the patient or ability to complete the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Clinical equivalence of ECG intervals compared between AIMIGo Synthesized 12L and reference standard 12L | 30 seconds recording
  Quantitative analysis on ECG intervals of the median beat of a 30s simultaneously recorded ECG from study and reference device.
Clinical equivalence of ECG amplitudes compared between AIMIGo Synthesized 12L and reference standard 12L | 30 seconds recording
  Quantitative analysis on ECG amplitudes of the median beat of a 30s simultaneously recorded ECG from study and reference device.

SECONDARY OUTCOMES:
Clinical diagnostic accuracy of AIMIGo Synthesized 12L compared with the reference standard 12L ECG for the classification of arrhythmia. | 30 seconds recording
  Summary statistics demonstrating agreement on arrhythmia diagnoses between the two devices will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Fitzgerald, MD, PhD, Study Director — HeartBeam, Inc.
Locations (5):
- United States (5):
  - Piedmont Heart Institute, Atlanta, Georgia
  - Atlanta Heart Specialists, Tucker, Georgia
  - The Mount Sinai Hospital, New York, New York
  - Long Island Jewish Medical Center, Queens, New York
  - Allegheny Health Network, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: HeartBeam Website — https://www.heartbeam.com/